CLINICAL TRIAL: NCT06446154
Title: Fruquintinib in Patients With Unresectable Hepatocellular Carcinoma Previously Treated With Immune Checkpoint Inhibitors : A Single-arm, Phase II Study
Brief Title: Fruquintinib After ICIs Treatment in Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRU-001
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; Immune Checkpoint Inhibitors; Anti-angiogenic Therapy; Second-line Treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — HMPL-013

STUDY DESIGN:
Intervention Model Description: Fruquintinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib (Experimental): Fruquintinib monotherapy
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib was given orally for 5mg/ days. After 3 weeks, the drug was stopped for 1 week.

SUMMARY:
Nowadays, there are few second-line treatment options for advanced hepatocellular carcinoma (HCC). In order to further improve the efficacy of second-line treatment for advanced HCC, we plan to conduct a phase II clinical study to explore the efficacy and safety of the new second-line treatment for advanced HCC.

As a tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor -1/2/3 (VEGFR 1/2/3), fruquintinib had demonstrated a strong antitumor efficacy in colorectal cancer patients who had previously received standard chemotherapy. Compared with placebo, fuquinitinib significantly extended overall survival in patients with metastatic colorectal cancer (median OS, 9.3 months vs 6.6 months; HR, 0.65; p<0.001) and progression-free survival (median PFS, 3.7 months vs 1.8 months; HR, 0.26; p<0.001). Additionally, a phase II clinical study had showed that sintilimab combined with fruquintinib was with a promising anti-tumor activity in patients with advanced HCC who had received standard treatment, with a median PFS of 7.4 months and a tumor response rate of 31.6%.

Therefore, we intend to conduct this clinical study to explore the efficacy and safety of fruquintinib as second-line treatment for patients with unresectable HCC previously treated with immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* with unresectable, locally advanced, or metastatic HCC, with the diagnosis confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Disease criteria
* who had previously received immune checkpoint inhibitors
* had at least on measurable disease, as defined by Response Evaluation Criteria In Solid Tumours version 1.1 (RECIST v1.1) criteria
* had a baseline Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* had a Child-Pugh liver function score of 7 or less
* had adequate hematologic and organ function (absolute neutrophil count ≥1.2×109/l, platelet count ≥60×109/l, total bilirubin < 30μmol/l, albumin ≥ 30g/l, aspartate transaminase and alanine transaminase ≤ 5×upper limit of the normal, creatinine clearance rate of ≤ 1.5×upper limit of the normal, and left ventricular ejection ≥ 45%)

Exclusion Criteria:

* history of HIV, organ allograft
* combined with other malignant tumors
* evidence of hepatic decompensation, bleeding diathesis or event
* allergy to the investigational agents or any agent given in association with this trial
* incomplete medical information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Two years
  Objective response rate

SECONDARY OUTCOMES:
OS | Two years
  Median overall survival
PFS | Two years
  Median progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No